CLINICAL TRIAL: NCT07266480
Title: A Randomised, Controlled Clinical Study of Adebrelizumab for the Adjuvant Treatment of Esophageal Squamous Cell Cancer.
Brief Title: Clinical Study of Adbelimumab in the Adjuvant Treatment of Esophageal Squamous Cell Carcinoma.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARL-ESCC
Record Dates: First submitted 2025-08-18; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-08

CONDITIONS: Squamous Oesophageal Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adebrelizumab (Experimental): Adebrelizumab: 1200mg, iv, d1, q3w, 17 cycles
  Interventions: Drug: Adebrelizumab
- close follow-up (No Intervention)

INTERVENTIONS:
Drug: Adebrelizumab — Patients undergoing radical surgery to achieve R0 resection were randomised in a 1:1 ratio at 4-16 weeks postoperatively, with patients in the trial group receiving adjuvant treatment with adebrelizumab (up to 17 cycles)
  Arms: Adebrelizumab

SUMMARY:
Evaluating the efficacy and safety of adebrelizumab for the adjuvant treatment of esophageal squamous cell cancer.

ELIGIBILITY:
Inclusion Criteria:

1.Age:≥18 years old, male or female; 2.Histopathologically confirmed esophageal squamous cell cancer with initial clinical stage cT1b-2N1-3M0 or cT3-4aN0-3M0 in the thoracic esophagus; 3.Radical surgery with R0 resection 4-16 weeks prior to randomisation; 4.Eastern Cooperative Oncology Group (ECOG) performance status of 0-1; 5.Expected survival ≥ 12 months; 6.Left ventricular ejection fraction is >50%; 7.Normal functioning of major organs, i.e. meeting the following criteria:

1. routine blood tests:

   1. HB≥90g/L；
   2. ANC≥1.5×109/L；
   3. PLT≥100×109/L；
2. biochemical examination:

   1. ALT and AST<2.5ULN（liver metastasis: ALT and AST<5ULN）；
   2. TBIL≤1.5ULN；
   3. creatinine ≤1.5ULN； 8.Participants were willing to join in this study, written informed consent, good adherence and co-operation with follow up.

Exclusion Criteria:

1. Patients initially diagnosed as unresectable (e.g. large metastatic lymph nodes) and treated with conversion therapy;
2. Patients with severe postoperative complications who are not suitable for adjuvant therapy;
3. Patients who have received any form of adjuvant therapy after surgery;
4. Patients who have received or are receiving other chemotherapy, radiotherapy or targeted therapy;
5. Pre-existing other malignancies, unless complete remission was achieved at least 5 years prior to enrolment and no other treatment is expected to be required during the study period;
6. Patients with active, known or suspected autoimmune disease, including but not limited to: interstitial pneumonitis, enteritis, hepatitis, pituitary gland inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism (may be considered for inclusion after hormone replacement therapy); patients with psoriasis or childhood asthma/allergies that have been in complete remission and do not require any intervention in adulthood may be considered for inclusion, but medical intervention with bronchodilator is required patients may not be included;
7. People with active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection;
8. Pregnant or breastfeeding women and women of childbearing age with a history of immunodeficiency, including HIV-positive, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation or allogeneic bone marrow transplantation who are not using contraception during the trial period;
9. Presence of clinically uncontrolled cardiac symptoms or disease, including but not limited to, such as (1) NYHA class II or higher heart failure, (2) unstable angina, (3) myocardial infarction within 6 months, (4) clinically significant supraventricular or ventricular arrhythmia not clinically intervened with or poorly controlled after clinical intervention;
10. Not suitable for enrolment in the investigator's comprehensive assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
DFS | 3 years
  DFS is defined as the time from registration to the first of the following events: local/regional ipsilateral invasive recurrence (or ipsilateral invasive new primary), contralateral invasive breast cancer, distant recurrence, or death from any cause. Patients without an event are censored at the date of last evaluation.

SECONDARY OUTCOMES:
OS | 3 years
  Baseline to measured date of death from any cause
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 3 years
  Through continuous monitoring and analysis of the safety data, the drug safety characteristics were evaluated, the suspected and unexpected serious adverse reactions and other major risks were identified in time, and appropriate measures were taken to fully control the risks and protect the safety of the subjects.
Patient reported outcome (Quality of Life questionnaire of cancer patients) | At the end of Cycle 1 (each cycle is 21 days)
  EORTC Quality of Life-Core 30/18 questionnaire module

CONTACTS AND LOCATIONS:
Locations (1):
- 12, Jiankang road, Chang'an District, Shijiazhuang, Hebei 050000, China, Shijiazhuang, Hebei, China